CLINICAL TRIAL: NCT06932523
Title: Randomized, Blinded, Controlled Phase I/Ⅱ Clinical Trial Evaluating the Safety and Immunogenicity of Recombinant Herpes Zoster Vaccine (CHO Cells) for Healthy Individuals Aged 40 Years and Above
Brief Title: A Study to Evaluate the Safety of Recombinant Herpes Zoster Vaccine for Healthy Individuals
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SIBP-V04-Ⅰ/Ⅱ
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Herpes Zoster (HZ)
Keywords: herpes zoster; recombinant herpes zoster vaccine; vaccine; safety; immunogenicity
MeSH Terms: conditions — Herpes Zoster | interventions — Adjuvants, Pharmaceutic; halofantrine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- SubStudy A (SSA): Group 1 (Experimental): Recombinant herpes zoster vaccine with low-dose adjuvant
  Interventions: Biological: Recombinant herpes zoster vaccine with low-dose adjuvant
- SSA: Group 2 (Experimental): Recombinant herpes zoster vaccine with high-dose adjuvant
  Interventions: Biological: Recombinant herpes zoster vaccine with high-dose adjuvant
- SSA:Control group 1 (Placebo Comparator): Low-dose adjuvant
  Interventions: Biological: Low-dose adjuvant
- SSA:Control group 2 (Placebo Comparator): High-dose adjuvant
  Interventions: Biological: High-dose adjuvant
- SSA: Positive control (Active Comparator): Shingrix (GSK)
  Interventions: Biological: Shingrix (GSK)
- SSA: Placebo group (Placebo Comparator): Normal saline
  Interventions: Biological: Normal Saline
- SubStudy B (SSB): Group 3 (Experimental): Recombinant herpes zoster vaccine with low-dose adjuvant
  Interventions: Biological: Recombinant herpes zoster vaccine with low-dose adjuvant
- SSB: Group 4 (Experimental): Recombinant herpes zoster vaccine with high-dose adjuvant
  Interventions: Biological: Recombinant herpes zoster vaccine with high-dose adjuvant
- SSB: Positive control (Active Comparator): Shingrix (GSK)
  Interventions: Biological: Shingrix (GSK)
- SSB: Placebo group (Placebo Comparator): Normal saline
  Interventions: Biological: Normal Saline

INTERVENTIONS:
Biological: Recombinant herpes zoster vaccine with low-dose adjuvant — Candidate 1, Dose Level 1, Intramuscular injection, 0, 2 months schedule
  Arms: SubStudy A (SSA): Group 1; SubStudy B (SSB): Group 3
Biological: Recombinant herpes zoster vaccine with high-dose adjuvant — Candidate 2, Dose Level 2, Intramuscular injection, 0, 2 months schedule
  Arms: SSA: Group 2; SSB: Group 4
Biological: Low-dose adjuvant — Adjuvant control 1, Dose Level 1, Intramuscular injection, 0, 2 months schedule
  Arms: SSA:Control group 1
Biological: High-dose adjuvant — Adjuvant control 2, Dose Level 2, Intramuscular injection, 0, 2 months schedule
  Arms: SSA:Control group 2
Biological: Shingrix (GSK) — Positive control, Intramuscular injection, 0, 2 months schedule
  Arms: SSA: Positive control; SSB: Positive control
Biological: Normal Saline — Placebo control, Intramuscular injection, 0, 2 months schedule
  Arms: SSA: Placebo group; SSB: Placebo group

SUMMARY:
The purpose of this clinical study is to evaluate the safety and immunogenicity of receiving two doses of recombinant herpes zoster vaccine (CHO cells) (RHZV) in healthy individuals aged 40 years and above. This study will be conducted in 2 substudies: Substudy A (Phase I) and Substudy B (Phase Ⅱ).

DETAILED DESCRIPTION:
There are two parts of the study.

Substudy A:

This substudy is the Phase I portion of the study. In this substudy, participants will receive 1 of 2 RHZV candidates (different dose levels) or the approved shingles vaccine (positive control) or adjuvant controls or normal saline intramuscularly. Participants will be divided into 2 age groups: 40-49 years old and ≥ 50 years old. Participants will receive vaccinations on days 0 and 60. Participants will complete a 12-month safety follow-up after two doses of vaccination, and they will take part in this study for about 14 months.

Substudy B:

This substudy is the Phase Ⅱ portion of the study. In this part of the study, participants will also receive 1 of 2 RHZV candidates (different dose levels) or the approved shingles vaccine (positive control) or normal saline intramuscularly. Participants will be divided into 3 age groups: 40-49 years old, 50-69 years old and ≥ 70 years old. Participants will receive vaccinations on days 0 and 60. Some group(s) will continue into persistence-of-immunity (overtime assessment of effect of vaccine) portion of the study. Those participants will be involved in this study for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years old on the day of enrollment, gender not limited.
* Can provide legal proof of identity.
* Be able to understand the experimental procedure and sign a written informed consent form, expressing agreement to participate in the experiment.
* Be able to participate in all planned follow-up visits and comply with all trial procedures.
* On the day of enrollment, the body temperature was less than 37.3 ℃ (axillary temperature).
* Chronic disease patients need to be in a stable period of chronic disease.
* Female and male participants of childbearing age agreed to adopt strict and effective contraceptive measures from the start of the trial to 6 months after full exemption.

Exclusion Criteria:

* Individuals with a history of herpes zoster in the past.
* Individuals with a history of vaccination against chickenpox or shingles.
* Individuals who have had close contact with patients with chickenpox or shingles in the past 2 years.
* Women of childbearing age who have a positive urine pregnancy test, are breastfeeding, pregnant, or plan to become pregnant within 6 months after the start of the test and the full exemption period.
* Individuals who are allergic to any component of the vaccine or have a history of other severe allergies.
* Use immunoglobulin and/or any blood products within 3 months prior to administering the trial vaccine, or plan to use them during the trial period.
* Have taken antipyretic, analgesic, or anti allergic drugs within 72 hours prior to receiving the experimental vaccine.
* Any experimental or unregistered product (drug, vaccine, biological product or device) other than the experimental vaccine has been used within one month prior to vaccination, or is planned to be used during the trial period.
* Administer non live vaccines within 7 days prior to administering the experimental vaccine or live vaccines within 14 days prior to administering the experimental vaccine.
* Suffering from a serious illness that prevents the completion of the entire experiment.
* Received immunosuppressive therapy or other immunomodulatory drugs, monoclonal antibodies, thymosin, interferon, etc. within 6 months prior to vaccination with the experimental vaccine, or planned to receive such treatment within 1 month after the first dose to full immunization, but local medication is allowed.
* Chemotherapy, radiotherapy, and organ and bone marrow transplantation related treatments for cancer or other diseases.
* Diseases or medical measures that lead to immune dysfunction
* Individuals currently suffering from serious infectious diseases such as active tuberculosis and active viral hepatitis.
* Moderate or severe acute illness/infection, or febrile illness within 72 hours prior to vaccination.
* Known to have a history of thrombocytopenia, any coagulation dysfunction, or being treated with anticoagulants.
* Suffering from serious cardiovascular disease, pulmonary edema, serious liver and kidney disease, and diabetes that cannot be controlled by drugs.
* Previous history of mental and neurological disorders or family history of mental illness.
* Currently suffering from various severe infectious, suppurative, and allergic skin diseases.
* Plan to move before the end of the trial or leave the local area for a long time during the scheduled trial visit.
* (Phase I ) Abnormal blood routine, blood biochemistry, coagulation, and urine routine indicators before vaccination (excluding those judged by doctors to have no clinical significance).
* Any situation that the researcher believes may affect the evaluation of the experiment.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 645 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of immediate Adverse Events (AEs) | 30min after each dose of vaccination
  The occurrence of any adverse events within 30 minutes after each dose of vaccination.
Percentage of solicited Adverse Events | 14 days after each dose of vaccination
  Adverse events defined by the protocol that occurred to the participant during 0-14 days after each dose of vaccination.
Serious Adverse Events (SAE) | 12 months after the last dose
  That is serious adverse events, any serious adverse events that occurred to the participant during the study period.
Percentage of unsolicited Adverse Events | 28 or 30 days after each dose of vaccination
  Other adverse events that occurred among participants within 0-28/30 days after each vaccination, in addition to the solicited adverse events.
Geometric Mean Concentration (GMC) of Anti-glycoprotein E (gE) Antibodies | 30 days after the last dose of vaccination
  GMC levels o of Anti-gE Antibodies in participants after receiving 2 doses of vaccine.
Geometric Mean Titer (GMT) of Anti-VZV Antibodies | 30 days after the last dose of vaccination
  GMT levels o of Anti-VZV Antibodies in participants after receiving 2 doses of vaccine.
Positive rate of Anti-gE Antibodies | 30 days after the last dose of vaccination
  The proportion of individuals in the study population who have achieved Anti-gE antibody positive after immunization.
Positive rate of Anti-VZV Antibodies | 30 days after the last dose of vaccination
  The proportion of individuals in the study population who have achieved Anti-VZV antibody positive after immunization.
Seroconversion rate of Anti-gE Antibodies | 30 days after the last dose of vaccination
  The proportion of individuals in the study population who have achieved Anti-gE antibody seroconversion after immunization.
Seroconversion rate of Anti-VZV Antibodies | 30 days after the last dose of vaccination
  The proportion of individuals in the study population who have achieved Anti-VZV antibody seroconversion after immunization.

SECONDARY OUTCOMES:
SSB： Cellular immune level | 30 days, 6 months, 12months and 24 months after the last dose of vaccination
  Levels of glycoprotein E (gE)-specific CD4+/CD8+ T cells expressing 2 or more markers of activation.
SSB：Humoral immunogenicity level | 6 months, 12months and 24 months after the last dose of vaccination
  Levels of GMC (Anti-gE antibody), GMT (Anti-VZV antibody), positive rate and seroconversion rate after receiving 2 doses of vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Yeqing Tong, Principal Investigator — Hubei Provincial Center for Disease Control and Prevention
Locations (1):
- Hubei Provincial Center for Disease Control and Prevention, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No